CLINICAL TRIAL: NCT03019211
Title: Feasibility of a Physical Exercise Program, Performed Inside or Outside the Aquatic Environment, to Reduce Falls in Institutionalized Elderly: A Pilot Randomised Clinical Study
Brief Title: Feasibility Aquatic Physical Exercise to Reduce Falls in Institutionalized Elderly
Acronym: PrePhysFalls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Collaborators: Sanitas Mayores Les Corts (Unknown); Residencial Augusta Park (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PrePhysFalls
Record Dates: First submitted 2017-01-08; First posted 2017-01-12 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2016-09

CONDITIONS: Age Problems; Cognitive Impairment; Elderly; Postural Balance; Strength
Keywords: Physical Therapy Modalities; Accidental Fall; Elderly; Hydrotherapy; Nursing Home
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrotherapy (Experimental): Exercise performed in an aquatic environment. The participants will perform static/dynamic exercises (balance and resistance training) in an aquatic environment. Training volume and intensity we will increase systematically over 12 weeks.
  Interventions: Other: Exercise
- Control (Active Comparator): The participants will perform exercises (balance and resistance training) like hydrotherapy group but out of the aquatic environment, during a 12 weeks training period (3sessions/week). Training volume and intensity we will increase systematically over 12 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
This is a pilot randomized control trial with single blinding of the assessor that will be conducted in two nursing homes residence to evaluate the applicability of a physical exercise program performed in an aquatic environment compared with the same realization but land-based to reduce falls in the institutionalized old people. The secondary objectives are to study the applicability of the intervention in improving balance, function, gait mobility, muscle strength of the lower limbs and the perception of the intervention.

DETAILED DESCRIPTION:
The participants will be randomized and divided into the hydrotherapy group or the control group. Each participant will attend a total of 24 physical exercise sessions of 50 minutes of duration. The study outcomes will be measured before the intervention and in 3 posterior phases to evaluate its effects in the short, medium and long terms.

ELIGIBILITY:
Inclusion Criteria:

* Be institutionalized in a care center
* Participate voluntarily and sign the informed consent
* Have a punctuation of 2 or more in The Downton Fall Risk Index

Exclusion Criteria:

* Suffer from a condition that can be affected or hinder exercise
* Acute disease unresolved in 10 days
* Not controlled hypertension
* Contagious skin disorder
* Urinary or faecal incontinence

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline Number of Falls at 3 months, 6 months and 9 months | 3 months, 6 months, 9 months
  Falls follow up

SECONDARY OUTCOMES:
Balance measured with Performance Oriented Mobility Assessment | 3 months, 6 months, 9 months
  Measured with Performance Oriented Mobility Assessment
Pain measured with Visual Analogue Scale | 3 months, 6 months, 9 months
  Measured with Visual Analogue Scale
Mobility measured with Timed Up & Go Test | 3 months, 6 months, 9 months
  Measured with Timed Up & Go Test
Daily living activities measured with Barthel Test | 3 months, 6 months, 9 months
  Measured with Barthel Test
Muscle strength measured with Five Sit to Stand test and Handgrip Test | 3 months, 6 months, 9 months
  Measured with Five Sit to Stand test and Handgrip Test
Intervention Perception measured with Qualitative interview | 3 months
  Qualitative interview

CONTACTS AND LOCATIONS:
Overall Officials: Mercè Sitjà Rabert, PhD, PT, Principal Investigator — University Ramon Llull
Locations (1):
- Universitat Ramon Llull, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No